CLINICAL TRIAL: NCT04034186
Title: The Assessment of the Content and Quality of Physiotherapy Management and Advice in Chronic Low-back Pain Patients in Central Finland
Brief Title: The Quality of Physiotherapy in Low Back Pain Patients in Central Finland
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Juhani Multanen (Other)
Responsible Party: Sponsor-Investigator, Juhani Multanen, Exercise physiologist, MSc, Central Finland Hospital District
Organization: Central Finland Hospital District (Other)
Other Study IDs: Dnro 2E/2014
Record Dates: First submitted 2015-08-17; First posted 2019-07-26 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2019-07

CONDITIONS: Low Back Pain
Keywords: low back pain; rehabilitation; assessment; quality
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic low back pain is one of the most common musculoskeletal disorders. In the Finnish Health 2000 survey the incidence of low back pain was 10% in men and 11% in women. Several evidence-based rehabilitation guidelines recommend exercise therapy treatment of chronic back pain. However, there are no studies in chronic low back pain patients concerning the assessment of the content and quality of exercise modalities adviced in clinical practise.

The aim of this study is to investigate the content and quality of physiotherapy management and advise in chronic low back pain patients in Central Finland.

DETAILED DESCRIPTION:
The participants in this study are 100 working-age unspecific low back pain patients from the Central Health Care District, who are referred for specialised care in the outpatient clinic in the Department of Physical Medicine and Rehabilitation in Central Finland Hospital. The participants will be asked to complete health-related questionnaires and an in-house made questionnaire of their back rehabilitation. The main questions are:

1. The content about applied exercise modalities,
2. How the progression of exercises have been advised?
3. How pain was taken into account while exercising? The research will be carried out and coordinated by Central Finland Central Hospital, and the research project will take place between November 2014 and February 2019.

ELIGIBILITY:
Inclusion Criteria:

* experiencing chronic low back pain,
* ability to communicate in Finnish language

Exclusion Criteria:

* previous back surgery in the preceding 12-month
* suspected or diagnosed lumbar disc herniation

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unspecified chronic (symtoms >12 weeks) low back pain referred to the outpatient clinic in the Department of Physical Medicine and Rehabilitation in Central Finland Hospital, Jyväskylä.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Self-constructed questionnaire; the content about instructed exercise modalities | During the physiotherapy treatment period
  Strength training, aerobic exercise, aquatic exercise, mobility or something else

SECONDARY OUTCOMES:
Self-constructed questionnaire; the way how the training was instructed by the physiotherapist | During the physiotherapy treatment period
  Verbally, in written form or by practicing
Self-constructed questionnaire; how back pain was taken into account in exercise guidance? | During the physiotherapy treatment period
  Patient did not receive instructions on how pain should be taken into account while exercising, patient was urged to avoid exercises that caused pain while exercising, patient was urged to exercise within the limits of pain, patient was urged to practice despite the pain, some other instructions - what?

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, Docent, Principal Investigator — Chief physician in the Department of Physical Medicine and Rehabilitation, Central Finland Central Hospital